CLINICAL TRIAL: NCT02265302
Title: A Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Investigate the Safety, Tolerability, Biological Effects and Preliminary Pharmacokinetics of Increasing Single Oral Doses of BIIL 284 BS (Dose Range: 0.025 mg - 75 mg PSE Solution, 25 mg, 75 mg, 250 mg and 750 mg WIF Tablets) in Healthy Male Volunteers as Well as Food Effects at 75 mg (WIF Tablet)
Brief Title: Safety, Tolerability, Biological Effects and Pharmacokinetics of BIIL 284 BS in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.1
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — amelubant; Tablets

ARMS (3):
- BIIL 284 BS oral solution (Experimental)
  Interventions: Drug: BIIL 284 oral solution
- BIIL 284 BS WIF tablets (Experimental)
  Interventions: Drug: BIIL 284 wetability improved formulation (WIF) tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 oral solution
  Arms: BIIL 284 BS oral solution
Drug: BIIL 284 wetability improved formulation (WIF) tablets
  Arms: BIIL 284 BS WIF tablets
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to obtain information about the safety and tolerability of BIIL 248 BS, to find the pharmacologically active dose range for the two formulations PSE 1% and WIF tablets by determination of the surrogate marker CD11b (= Mac-1) and to obtain preliminary pharmacokinetic data as well as first information on food effects after administration of the 75 mg WIF tablet in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Age ≥ 21 and ≤ 50 years
* Broca ≥ - 20% and ≤ + 20%
* Signed written informed consent in accordance with Good Clinical Practice and local legislation

Exclusion Criteria:

* Results of the medical examination or laboratory tests that are judged by the clinical investigator to differ significantly from normal clinical values
* Known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Known history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (≥ 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Intake of any other drugs which might influence the results of the trial during the week previous to the start of the study
* Participation in another study with an investigational drug within the last two months preceding this study
* Smokers (> 5 cigarettes or 2 cigars or 2 pipes/day)
* Volunteer who is not able to refrain from smoking on study days
* Alcohol abuse (more than 60 g of alcohol per day)
* Drug abuse
* Excessive physical activities (e.g. competitive sports) within the last week before the study
* Blood donation within the last 4 weeks (≥ 100 ml)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 1998-06; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically relevant changes in vital signs | up to 8 days after drug administration
Number of subjects with clinically relevant changes in electrocardiogram | up to 8 days after drug administration
Number of subjects with clinically relevant changes in laboratory parameters | up to 8 days after drug administration
Number of subjects with adverse events | up to 8 days after drug administration
Determination of surrogate marker cluster of differentiation antigen 11b (CD11b) (=Mac-1) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Changes in white blood cell count | up to 48 hours after drug administration
  determined by flow cytometer
Changes in differential blood cell count | up to 48 hours after drug administration
  determined by flow cytometer
Maximum plasma concentration (Cmax) | up to 72 hours after drug administration
Time to reach maximum plasma concentration (tmax) | up to 72 hours after drug administration
Area under the plasma concentration-time curve (AUC) for several time intervals | up to 72 hours after drug administration
Terminal half-life (t1/2) | up to 72 hours after drug administration
Total mean residence time (MRTtot) | up to 72 hours after drug administration
Total clearance after oral administration (CLtot/f) | up to 72 hours after drug administration
Volume of distribution during terminal phase after oral administration (Vz/f) | up to 72 hours after drug administration